CLINICAL TRIAL: NCT03947606
Title: An Optimization Trial to Prepare Advanced Cancer Caregivers for Decision Partnering Using the Multiphase Optimization Strategy (MOST)
Brief Title: Pilot Optimization Trial of Decision Partnering Intervention for Advanced Cancer Family Caregivers
Acronym: CASCADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, James N Dionne-Odom, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-#300003601
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Family Caregivers; Cancer
Keywords: Decision-making; Decisions; Multiphase Optimization Strategy; Factorial design
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: 2x2x2 full factorial pilot randomized trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data collectors and principal investigator will be blind to participant condition; participants will be instructed NOT to discuss their assignment with data collectors. Trials participants will know their intervention condition as will the nurse coach involved in delivering the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Basic social support + communication + Ottawa guide (Experimental): 3 in-person/telephone weekly sessions on providing decision social support, tips for good communication, and decision support tools
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Basic social support + communication (Experimental): 2 in-person/telephone weekly sessions on providing decision social support and tips for good communication
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Basic social support + Ottawa guide (Experimental): 2 in-person/telephone weekly sessions on providing decision social support and decision support tools
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Basic social support only (Experimental): 1 in-person/telephone weekly session on providing decision social support
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Advanced social support + communication + Ottawa guide (Experimental): 5 in-person/telephone weekly sessions on providing decision social support, tips for good communication, and decision support tools
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Advanced social support + communication (Experimental): 4 in-person/telephone weekly sessions on providing decision social support and tips for good communication
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Advanced social support + Ottawa guide (Experimental): 4 in-person/telephone weekly sessions on providing decision social support and decision support tools
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)
- Advanced social support only (Experimental): 3 in-person/telephone weekly sessions on providing decision social support
  Interventions: Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners)

INTERVENTIONS:
Behavioral: CASCADE (CAre Supporters Coached to be Adept DEcision partners) — CASCADE (CAre Supporters Coached to be Adept DEcision partners) is a multicomponent, nurse coach-led supportive care intervention designed to increase family caregivers' skills in providing decision support to individuals with advanced cancer. In a series of weekly, one-on-one, 15-20 minute, in-person or telephone sessions, family caregivers receive psychoeducation on principles of providing effective social support and decision partnering, decision support communication, and Ottawa Decision Guide training.

SUMMARY:
Using a highly innovative methodology, the Multiphase Optimization Strategy (MOST), the purpose of this study is to pilot test, for the first time, an optimization trial approach to develop and refine the decision partnering skills of family caregivers of persons with newly-diagnosed advanced cancer. Using a 2x2x2 full factorial design, 40 family caregivers of persons with newly-diagnosed advanced cancer will be randomized to receive one or more nurse coach-delivered decision partnering training components, based on the Ottawa Decision Support Framework and Social Support Effectiveness Theory4: 1) psychoeducation on effective decision partnering principles (1 vs. 3 sessions); 2) decision partnering communication training (yes vs. no); and 3) Ottawa Decision Guide training (yes vs. no).

DETAILED DESCRIPTION:
A priority focus in palliative care, oncology, and geriatrics is preparing the 2.8 million U.S. family caregivers of persons with cancer to effectively partner with patients in healthcare decision-making from diagnosis to the end of life. Over 70% of patients with cancer report involvement by relatives, friends, and partners in healthcare decisions, including choices about cancer treatments, surgery, transitions and location of care, accessing palliative and hospice care, and many others. Hence, there is a critical need to train cancer family caregivers to be supportive of patient decision-making; however, few palliative care interventions exist that enhance skills in effective decision partnering. Patients making healthcare decisions with unprepared family caregivers may experience inadequate family decision support leading to heightened distress and receipt of care/treatments inconsistent with their values and preferences. This in turn may increase distress for family caregivers.

Becoming better decision partners with patients is one among several skills targeted within our evidence-based model of early concurrent oncology palliative care for family caregivers. Decision partnering relevant content for family caregivers has included principles of effective social support, communication, and Ottawa Decision Guide training; however it is unknown which of these components and component interactions influences patient and caregiver decision-making outcomes. Traditional research approaches typically treat interventions as "bundled" treatment packages, making it difficult to assess definitively which aspects of an intervention can be reduced, eliminated, or replaced to improve efficiency. Using traditional research methods (e.g., two-arm randomized controlled trials that test new features one at a time) requires conducting multiple studies, which is an exorbitantly expensive and time consuming process. This paradox prompts us to consider methodologies that may offer a more efficient way to test multiple intervention components simultaneously.

Using a highly innovative methodology, the Multiphase Optimization Strategy (MOST), the purpose of this study is to pilot test, for the first time, an optimization trial approach to develop and refine the decision partnering skills of family caregivers of persons with newly-diagnosed advanced cancer (CASCADE: CAre Supporters Coached to be Adept DEcision partners). Using a 2x2x2 factorial design, 40 family caregivers of persons with newly-diagnosed advanced cancer will be randomized to receive one or more nurse coach-delivered decision partnering training components, based on the Ottawa Decision Support Framework and Social Support Effectiveness Theory4: 1) psychoeducation on effective decision partnering and social support principles (1 vs. 3 sessions); 2) decision support communication training (yes vs. no); and 3) Ottawa Decision Guide training (yes vs. no).

This study's conceptual foundations incorporate Rini's Social Support Effectiveness Theory and the Ottawa Decision Support Framework. Caregiver decision partnering training is designed to modify family caregiver skills, including their ability to: 1) provide effective social support through psychoeducation on key social support principles that will optimize emotional and informational support to patients; 2) elicit patient decisional needs, including patient values, preferences, and coping through better decision support communication, enhancing the quantity of decision-making conversations; and 3) provide structured decision support using an evidence-based tool (i.e., the Ottawa Decision Guide, see Appendix) to help patients clarify choices and guide deliberation through Ottawa decision guide training, reducing patient decision conflict. Modification of these skills and improvement in patient mediating outcomes is hypothesized to lead to more positive decisional influence from the patient's perspective and better patient and caregiver mood.

The specific aims of this study are to:

Aim 1: Determine the feasibility and acceptability of using a highly innovative experimental design to enroll and retain 40 caregivers for 24 weeks to complete 1 or more components of caregiver decision partnering training. Feasibility: ≥80% of participants will adhere to and complete assigned intervention components and study-related assessments. Acceptability: Through post-intervention qualitative interviews, the investigators will elicit feedback from caregiver participants on intervention experiences and clinical trial procedures.

Aim 2: Explore the preliminary efficacy of individual decision partnering training components and component interactions on patient and caregiver outcomes at 12 and 24 weeks after baseline, including a) patient-reported positive decision influence (primary) using Rini's Decision Influence Scale and b) patient and caregiver mood (depression/anxiety symptoms) using the Hospital Anxiety and Depression Scale.

Exploratory Aim: Explore mediators and moderators (e.g., sociodemographics, coping, social support, decisional conflict) of the relationship between intervention components and patient and caregiver outcomes.

ELIGIBILITY:
FAMILY CAREGIVERS

Inclusion:

1. ≥18 years of age;
2. Self-endorsing or identified by the patient as "a relative, friend, or partner that has a close relationship with you and who assists you with your medical decisions and who may or may not live in the same residence as you and who is not paid for their help";
3. Caring for a patient with advanced-stage cancer (see definition under Patient Inclusion criteria below);
4. Caregivers will need to have an agreeable patient willing to participate in the study (for data collection only);
5. English-speaking and able to complete baseline measures; and
6. Stated willingness to comply with all study procedures and be available for the duration of the study.

Exclusion:

1) Self-reported active severe mental illness (i.e., schizophrenia, bipolar disorder, or major depressive disorder), dementia, active suicidal ideation, uncorrected hearing loss, or active substance abuse

PATIENTS

Inclusion:

1. ≥18 years of age;
2. Diagnosed within past 60-90 days of initial pre-screening with an advanced cancer, defined as metastatic and/or recurrent/progressive stage III/IV cancer, including brain, lung, breast, gynecologic, head and neck, gastrointestinal, genitourinary cancer, melanoma; and hematologic malignancies;
3. English-speaking and able to complete baseline measures; and
4. Stated willingness to comply with all study procedures and be available for the duration of the study.

Exclusion:

1) Medical record documentation of active severe mental illness (i.e., schizophrenia, bipolar disorder, or major depressive disorder), dementia, active suicidal ideation, uncorrected hearing loss, or active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility | Baseline to 24 weeks
  Proportion of caregiver participants who complete assigned intervention components and proportion of caregiver and patient participants who complete study-related assessments.
Acceptability | Baseline to 24 weeks
  Through qualitative interviews, caregiver participant reported experiences with the CASCADE intervention and trial procedures.

SECONDARY OUTCOMES:
Patient-reported positive decision influence using Rini's Decision Influence Scale | 12 and 24 weeks after baseline
  30 items; assesses satisfaction with how family caregivers assist patient's with healthcare decision-making, such as acting angry, questioning or doubting the patient's decisions, failing to assist, making useful suggestions, listening, and offering helpful advice. Total score range: 37-185; higher scores=more positive decision influence by family member.
Patient mood using the Hospital Anxiety and Depression Scale | 12 and 24 weeks after baseline
  14 items; measures symptoms of anxiousness and depressed mood. 7 items measure anxiety (e.g., feeling tense, restless, worried) and 7 items measure depressive symptoms (e.g., cheerfulness, feeling slowed down. Subscale score ranges: 0-21; higher scores=worse anxiety or depressive symptoms. Total score range: 0-42; higher scores=worse overall distress.
Caregiver mood using the Hospital Anxiety and Depression Scale | 12 and 24 weeks after baseline
  14 items; measures symptoms of anxiousness and depressed mood. 7 items measure anxiety (e.g., feeling tense, restless, worried) and 7 items measure depressive symptoms (e.g., cheerfulness, feeling slowed down. Subscale score ranges: 0-21; higher scores=worse anxiety or depressive symptoms. Total score range: 0-42; higher scores=worse overall distress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No